CLINICAL TRIAL: NCT07224581
Title: A Multinational, Multicenter Study With an Open-Label Phase 1b and a Randomized, Double-Blind, Placebo-Controlled Phase 3 Followed by an Open-Label Extension to Assess the Efficacy, Safety, Tolerability, and Pharmacokinetics of Radiprodil in Participants With GRIN-Related Neurodevelopmental Disorder
Brief Title: Beeline: A Phase 3 Study in GRIN-related Neurodevelopmental Disorder
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GRIN Therapeutics, Inc. (Industry)
Collaborators: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Beeline RAD-GRIN-101
Record Dates: First submitted 2025-10-31; First posted 2025-11-04 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: GRIN-related Neurodevelopmental Disorder
Keywords: Beeline; GRIN1; GRIN2A; GRIN2B; GRIN2D; GRIN-NDD
MeSH Terms: interventions — radiprodil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: study personnel, sponsor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Radiprodil (Experimental): Liquid suspension of radiprodil, at varying concentrations depending on participant's weight.
  The following dose-escalation regimen (twice daily [BID]) will be used:
  Titration Period Visit 1 (Visit T1): Dose 1, Visit T2: Dose 2, Visit T3: Dose 3, Visit T4: Maintenance Dose.
  Interventions: Drug: Radiprodil
- Placebo (Placebo Comparator): Liquid suspension of placebo matching radiprodil oral suspension and dose-escalation regimen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Radiprodil — Radiprodil oral suspension
  Arms: Radiprodil
Drug: Placebo — Placebo-to-match radiprodil oral suspension
  Arms: Placebo

SUMMARY:
The Phase 3 portion of Study RAD-GRIN-101 is a multinational, multicenter, randomized, double-blind, placebo-controlled trial followed by an open-label extension to evaluate the efficacy and safety of radiprodil in participants with GRIN-related neurodevelopmental disorder (GRIN-NDD) with a gain-of-function (GoF) genetic variant.

This study will enroll two cohorts: one cohort of participants with a minimal number of countable motor seizures (with or without behavioral symptoms) (Phase 3 Cohort 1: Qualifying Seizures Cohort); and a second cohort with disease symptoms but no seizures or fewer seizures than required for the Qualifying Seizures Cohort (Phase 3 Cohort 2: Without Qualifying Seizures Auxiliary Cohort).

Participants in each cohort will be randomized 1:1 to receive active drug (radiprodil) or matching placebo (Part A). Following completion of Part A, all eligible participants (including those previously on placebo) may continue into the open-label extension period (Part B) to receive radiprodil.

The placebo-controlled portion is expected to be approximately 16 weeks for participants in Phase 3 Cohort 1 and 28 weeks for participants in Phase 3 Cohort 2.

The study will evaluate the effect of radiprodil on seizures and non-seizure symptoms and assess safety.

DETAILED DESCRIPTION:
Participants are assigned in a 1:1 ratio to receive either radiprodil or placebo during Part A with the opportunity to receive radiprodil in the Open-Label Extension, Part B. The dosing regimen includes a fixed titration schedule over 4 weeks.

This study is divided into the following parts:

Part A: Randomized, double-blind, placebo-controlled

* Screening/Observation Period: To assess eligibility
* Titration Period (approximately 4 weeks): Titration of radiprodil or placebo to target dose
* Maintenance Period (Part A): Target dose of radiprodil or placebo maintained for 12 weeks (Phase 3 Cohort 1) or 24 weeks (Phase 3 Cohort 2)
* Tapering and Follow-up Period: Gradual decrease and Follow-up Period for participants not entering Part B

Part B: Open-label safety follow-up period

* Open-Label Treatment Period: Participants will continue to receive radiprodil until such time as either the participant withdraws/is withdrawn from the study, sponsor terminates the study, or market access is available
* Tapering and Follow-up Period: Gradual decrease and follow-up observation period for participants upon leaving the study

ELIGIBILITY:
Inclusion Criteria:

Part A, Participant:

* Diagnosed with GRIN-NDD with GRIN1, GRIN2A, GRIN2B, or GRIN2D gene variants known to result in GoF of the NMDA receptor
* Phase 3 Cohort 1 (Qualifying Seizures Cohort) ONLY: Experiencing at least 1 CMS per week and ≥4 CMS (generalized or focal) during screening
* With history of inadequate response to at least 2 standard antiseizure medications (ASMs)
* Phase 3 Cohort 2 (Without Qualifying Seizures Auxiliary Cohort) ONLY: With significant neurodevelopmental symptoms and a GRIN-CGI-S score ≥4
* On a stable dose of standard ASMs for at least 4 weeks prior to screening and should remain on stable doses throughout study participation
* On stable nonpharmacological treatments such as ketogenic diet and should remain stable throughout study participation

Part B:

- Participant has completed Part A and is eligible to continue study participation according to the judgement of the investigator and sponsor.

Exclusion Criteria:

PART A, Participant:

* Has clinically relevant medical, neurologic, or psychiatric condition and/or behavioral disorder (including those related to GRIN-NDD) that would preclude or jeopardize participant's safe participation or study drug administration or the conduct of the study according to the judgement of the investigator or sponsor.
* Is receiving >4 standard ASMs at screening
* Has a body weight of less than 5 kg at screening

Part B:

- Participant has clinically relevant medical, neurologic, or psychiatric condition and/or behavioral disorder (including those related to GRIN-NDD) that would preclude or jeopardize participant's safe participation of study drug administration or the conduct of the study according to the judgement of the investigator or sponsor.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Part A - Phase 3 Cohort 1 (Qualifying Seizures Cohort): Countable motor seizures (CMS) | 12 weeks
Part A - Phase 3 Cohort 2 (Without Qualifying Seizures Auxiliary Cohort): Adverse events (AEs), serious adverse events (SAEs), and adverse drug reactions (ADRs) | 24 weeks
Part B - Open-Label Extension: Adverse events (AEs), serious adverse events (SAEs), and adverse drug reactions (ADRs) | Average of 2 years

SECONDARY OUTCOMES:
Part A - Phase 3 Cohort 1 (Qualifying Seizures Cohort): Proportion of participants with ≥50% reduction in CMS | 12 weeks
Part A - Phase 3 Cohort 1 (Qualifying Seizures Cohort): CMS-free days | 12 weeks
Part A - Phase 3 Cohort 1 (Qualifying Seizures Cohort): GRIN-NDD-specific Clinical Global Impression - Change [CGI-C] scale | 12 weeks
Part A - Phase 3 Cohort 1 (Qualifying Seizures Cohort): Aberrant Behavior Checklist-Community (ABC-2C) irritability subscale | 12 weeks
Part A - Phase 3 Cohort 1 (Qualifying Seizures Cohort): Vineland Adaptive Behavior Scale 3rd edition (VABS-3) daily living personal subdomain | 12 weeks
Part A - Phase 3 Cohort 2 (Without Qualifying Seizures Auxiliary Cohort): GRIN-CGI-C scale | 24 weeks
Part A - Phase 3 Cohort 2 (Without Qualifying Seizures Auxiliary Cohort): ABC-2C irritability subscale | 24 weeks
Part A - Phase 3 Cohort 2 (Without Qualifying Seizures Auxiliary Cohort): VABS-3 daily living personal subdomain | 24 weeks
PART B - Open-Label Extension: CMS frequency | average of 2 years
PART B - Open-Label Extension: CMS-free days | average of 2 years
PART B - Open-Label Extension: ABC-2C irritability subscale | average of 2 years
PART B - Open-Label Extension: VABS-3 daily living personal subdomain score | average of 2 years
PART B - Open-Label Extension: GRIN-CGI-C scale | average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alex Cepeda, Study Director — GRIN Therapeutics, Inc.; Russel Chin, Study Director — GRIN Therapeutics, Inc.
Locations (20):
- United States (20):
  - UCLA Health-Ronald Reagan Medical Center, Los Angeles, California
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Children's Hospital Colorado - Anschutz Medical Campus, Aurora, Colorado
  - Children's National Hospital, Washington D.C., District of Columbia
  - Nicklaus Children's Hospital, Miami, Florida
  - Pediatric Neurology and Epilepsy, Winter Park, Florida
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Northeast Regional Epilepsy Group (NEREG) - Hackensack, Hackensack, New Jersey
  - Columbia University - Harkness, New York, New York
  - Duke Health-Duke Children's Hospital & Health Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Child Neurology Consultants of Austin - South Austin, Austin, Texas
  - The University of Texas Southwestern Medical Center (UTSW), Dallas, Texas
  - UTHealth Houston, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided